CLINICAL TRIAL: NCT05205785
Title: Supporting Healthy Gastrointestinal Function With Human Milk Oligosaccharides (HMOs) in Individuals With Irritable Bowel Syndrome (IBS)
Brief Title: Human Milk Oligosaccharides (HMOs) for Irritable Bowel Syndrome (IBS)
Acronym: HIBS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to low enrollment, we have terminated this study
Sponsor: DSM Nutritional Products, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2021-07-21-HMOS
Record Dates: First submitted 2021-12-22; First posted 2022-01-25 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Irritable Bowel Syndrome; IBS - Irritable Bowel Syndrome
Keywords: Human Milk Oligosaccharides; HMOs
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Human Milk Oligosaccharide (HMO) mix (Experimental): The HMO blend to be used in this trial is a mix of the three milk oligosaccharides produced by fermentation of lactose. The blend is provided as white powder and mixed in a single serve stick packs containing 5.5 g of HMOs. The final product contains less than 0.03 g lactose per serving. The participants will be instructed to mix the product in a 4-6 oz glass of water and consume in the morning once a day for 12 weeks.
  Interventions: Dietary Supplement: Human Milk Oligosaccharide Mix
- Placebo (Placebo Comparator): The placebo to be used in this trial is 5.5 g of powdered dextrose powder in a single-serve stick pack. The participants will be instructed to mix the product in a 4-6 oz glass of water and consume in the morning once a day for 12 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Human Milk Oligosaccharide Mix — Subjects takes 5.5 g of powder mixed in water once a day for 12 weeks.
  Other Names: HMOs
  Arms: Human Milk Oligosaccharide (HMO) mix
Other: Placebo — The placebo to be used in this trial is 5.5 g of powdered dextrose powder in a single-serve stick pack. The participants will be instructed to mix the product in a 4-6 oz glass of water and consume in the morning once a day for 12 weeks.
  Arms: Placebo

SUMMARY:
To assess the effects of a Human Milk Oligosaccharide mix given once daily for 12 weeks on stool consistency and abdominal pain compared to placebo in individuals with Irritable Bowel Syndrome (IBS).

DETAILED DESCRIPTION:
HMO mix has been shown to provide therapeutic benefits to individuals with IBS of all subtypes (Palsson et al., 2019). DSM is planning this trial in order to investigate if clinically relevant improvements in bowel movements and IBS symptoms can be obtained through the use of the HMO mix in individuals with moderate to severe IBS and abdominal pain.

Eligible participants will have a diagnosis of Irritable Bowel Syndrome (IBS). Participants will be assessed for eligibility at the screening visit, must meet all the inclusion criteria, and none of the exclusion criteria.

In this trial, participants will be randomized to one of two intervention groups (a Human Milk Oligosaccharide mix or placebo) and receive intervention for at least 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained before any trial related assessments are performed.
2. Male or female aged ≥18 years at the time of consent.

   a. Female participants of child-bearing potential (females who are post-menopausal, i.e., when there has been no menstruation for a minimum of 12 months prior to screening, are considered not to be of child-bearing potential.), who are not surgically sterilized, must have a negative pregnancy test at screening and be willing to practice one of the following appropriate contraceptive methods until the last visit: i. Sexual abstinence. ii. Oral contraceptives. iii. Trans dermal patches or depot injection of a progestogen drug (starting at least 4 weeks prior to product administration). iv. Double barrier method: condom or occlusive cap (diaphragm or cervical/vault caps) plus spermicidal agent. v. Intrauterine device (IUD), intrauterine system (IUS), subdermal implant, or vaginal ring (placed at least 4 weeks prior to product administration). vi. Contraceptives must be effective before the randomization visit. However, national requirements should always be followed.
3. IBS-D or IBS-C or IBS-M according to Rome IV criteria. This will be established by using the IBS Module of the Rome IV Diagnostic Questionnaire, and requires recurrent abdominal pain on average at least 1 day per week during the previous 3 months that is associated with two or more of the following:

   1. Related to defecation (may be increased or unchanged by defecation) on at least 30% of pain instances in past 3 months.
   2. Associated with a change in stool frequency (on at least 30% of pain instances in past 3 months).
   3. Associated with a change in stool form or appearance (on at least 30% of pain instances in past 3 months).
4. Reported IBS diagnosis from a physician.
5. Personal access to the internet via computer, tablet, or smart-phone.
6. Be willing and able to comply with trial protocol, including entry of electronic diary data for at least 12 out of 14 diary days during the pre-randomization baseline 2-week run-in diary period (between V1 andV2).

   Inclusion criteria Visit 2: To be eligible for inclusion, the participant must fulfil all of the following criteria:
7. Scores of 1, 2, 6, or 7 on the Bristol stool scale at least twice per week [as determined by eDiary completion between V1 and V2].
8. An average baseline of worst abdominal pain of ≥3.3 (NRS-11) during the 2-week run-in period prior to randomization [as determined by eDiary completion between V1 and V2].

Exclusion Criteria:

The presence of any of the following criteria will exclude the participant from participating in the trial:

1. Treatment with an investigational drug from another clinical trial within 30 days/5 half- lives of the drug (which ever longest) prior to screening visit.
2. Any known gastrointestinal disease(s) or medical history that may interfere with the trial evaluations in the opinion of the investigator, in particular:

   1. Coeliac disease.
   2. IBD.
   3. Diverticulitis.
   4. C. difficile infection reported in the previous 2 years.
   5. Any clinically symptomatic biochemical or structural abnormality or active disease of the gastrointestinal tract within 6 months before screening, including daily diarrhea within two weeks prior to the screening interview or during the screening/baseline period.
   6. Substance abuse (within past 2 years).
   7. New use of antibiotics (within past 2 months), prebiotics, probiotics, or fiber supplements (within the past month).
   8. Hepatic dysfunction assessed as part of the blood safety panel (defined as alanine aminotransaminase/serum glutamic-pyruvic transaminase or aspartate aminotransaminase/serum glutamic-oxaloacetic transaminase >2.5 x the upper limit of normal, or a history of hepatobiliary disease) or renal impairment (serum creatinine) >2 mg/dl); any surgery (within a year of screening) on the stomach, small intestine, or colon (excluding appendectomy, hernia surgery not involving the GI tract, or c-section).
   9. Any history of pancreatitis (either acute or chronic).
   10. Laxative abuse (use of more than recommended dosage).
   11. Pregnant or lactating individuals.
   12. Any other gastrointestinal disease(s) or medical history that may interfere with the trial evaluations in the judgment of the investigator.
3. Following strict diets to improve their IBS symptoms as judged by the investigator e.g., Low FODMAP (within past 2 months). Exclusion based on diet will be reviewed by single investigator for consistency.
4. Any clinically relevant chronic disease(s) such as malignancy, diabetes, severe coronary disease, kidney disease, autoimmune or neurological disease, that in the opinion of the investigator would interfere with the trial evaluations or the safety of the participant.
5. Current severe psychiatric disease and/or psychological disturbance, a major psychiatric disorder requiring hospitalization in the last 3 years, or a history of attempted suicide or uncontrolled bipolar disorder; or clinical evidence of any significant psychiatric disease or symptoms that may interfere with the participant successfully completing the trial.
6. Treatment with restricted and prohibited concomitant medications.
7. Diagnosed with and treated for IBS for more than 10 years
8. Has a business or personal relationship with trial staff or sponsor who is directly involved with the conduct of the trial.
9. Lack of suitability for participation in the study for any reason as judged by the investigator.
10. Has previously been randomized into this trial, is participating in this trial at another investigational site or is planning to participate in any other clinical trial during this trial.
11. Desire and/or plans on changing current diet regime during the participation of this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2023-03-22 (Actual); Primary Completion 2024-03-05 (Actual); Study Completion 2024-06-24 (Actual)

PRIMARY OUTCOMES:
Absolute change in the proportion of stools with abnormal fecal consistency in the active product compared to placebo group. | Baseline (2 week run in period) to end of intervention (weeks 11 + week 12)
  Participants will identify each bowel movement 'type' using the Bristol Stool Scale (Type 1 = hard stool difficult to pass [classified as severe constipation]; Type 7 = watery, entirely liquid stool [classified as severe diarrhea]). Types 1 and 2 would be considered to suggest severe and mild diarrhea, respectively. Types 6 and 7 would be considered to suggest mild and severe diarrhea, respectively. This endpoint will compare the proportion of participants experiencing constipation and diarrhea between the groups
Absolute change in the pain severity score (IBS-SSS) in the active product compared to placebo group. | Baseline (Visit 2) to Week 12 (Visit 3)
  The IBS Symptom Severity Scale (IBS-SSS) contains a pain subscale which asks participants to rate abdominal pain the past 10 days on a scale from 0 to 100, with 0 meaning "no pain" and 100 meaning "very severe pain". The minimum score is 0 and the maximum achievable score is 100.

SECONDARY OUTCOMES:
Absolute change in total IBS severity score in the active product compared to placebo group. | Baseline (Visit 2) to Week 12 (Visit 3)
  The IBS Symptom Severity Scale (IBS-SSS) contains 5 items. Each of the five questions generate a maximum score of 100 using prompted visual analogue scales. The minimum score is 0 and the maximum achievable score is 500.
Absolute change in total IBS Quality of Life (IBS-QOL) score in the active product compared to placebo group. | Baseline (Visit 2) to Week 12 (Visit 3)
  The IBS Quality of Life contains 34 items each with a five-point response scale, where 1 represents not at all and 5 extremely/A great detail. The participant ill answer each question with respect to the impact of IBS and it's treatment. The individual responses to the 34 items are summed and averaged for a total score and transformed to a 0-100 scale for interpretation with higher scores indicating better IBS specific quality of life.
Relative change in abundance of fecal Bifidobacteria spp in the active product compared to placebo group. | Baseline (Visit 2) to Week 12 (Visit 3)
  Relative change in abundance measured by gene sequencing analysis of fecal sample.

OTHER OUTCOMES:
Absolute change in GSRS-IBS (Gastrointestinal Symptom Rating Scale-IBS) scores. | Baseline (Visit 2) to Week 12 (Visit 3)
  The Gastrointestinal Symptom Rating Scale- Irritable Bowel Syndrome questionnaire contains 13 items, each uses a seven-graded Likert scale, where 1 represents the most positive option (no symptoms) and 7 the most negative one (severe symptoms). The participant will answer each question with respect to their experience over the last 7 days. To calculate the Total Score, each of the 13 item scores will be used to calculate a mean Total Score: minimum possible score = 0; maximum possible score = 7; higher scores indicate worse symptoms.
  A mean value for the items in each dimension (Diarrhea; Constipation; Bloating; Pain & Satiety) will be calculated: minimum possible score = 0; maximum possible score = 7; higher scores indicate worse symptoms.
Abdominal pain responder rate. | Baseline (2-week run-in period) to the last two weeks of intervention (week 11+12)
  Based on the proportion of participants with a decrease in weekly average of worst abdominal pain of at least 30%.
Absolute change in BSFS (Bristol Stool Form Scale) score. | Baseline (2-week run-in period) to the last two weeks of intervention (week 11+12)
  Participants will identify each bowel movement 'type' using the Bristol Stool Scale (Type 1 = hard stool difficult to pass [classified as severe constipation]; Type 7 = watery, entirely liquid stool [classified as severe diarrhea]). Lower scores are indicative of constipation, and higher scores are indicative of diarrhea.
Absolute change in the number (or frequency) of bowel movements. | Baseline (2-week run-in period) to the last two weeks of intervention (week 11+12)
  Participants will report number of daily bowel movements. This endpoint will compare the change in number of bowel movements from baseline to end of intervention.
Percentage of participants with a decrease of 50 points in total IBS-SSS score. | Baseline (Visit 2) to Week 12 (Visit 3)
  The IBS Symptom Severity Scale (IBS-SSS) contains 5 items. Each of the five questions generate a maximum score of 100 using prompted visual analogue scales. The maximum achievable score is 500 with a decrease in score indicating a decrease in the severity of symptoms.
Absolute change in GAD-7 score. | Baseline (Visit 2) to Week 12 (Visit 3)
  The General Anxiety Disorder 7-item questionnaire (GAD-7) is a 7 item scale, each uses a four-graded Likert scale, where 0 represents the 'not at all' and 3 represents 'nearly every day'. The maximum score is 21 and scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively.
Absolute change in PHQ-8 score. | Baseline (Visit 2) to Week 12 (Visit 3)
  The Patient Health Questionnaire 8 (PHQ-8) is an 8 item scale. Each uses a four-graded Likert scale, where 0 represents 'not at all' and 3 represents 'nearly every day' and asks the participant how often (over the past two weeks) they have been bothered by each item. A total score of 0 to 4 represents no significant depressive symptoms; 5 to 9 represents mild depressive symptoms; 10 to 14, moderate symptoms; 15 to 19, moderately severe symptoms; and 20 to 24, severe symptoms.
Absolute change in WPAI-IBS (Work Productivity and Activity Impairment-IBS) score. | Baseline (Visit 2) to Week 12 (Visit 3)
  Absolute change measured by the WPAI-IBS.
Absolute change in BIPQ score. | Baseline (Visit 2) to Week 12 (Visit 3)
  The Brief Illness Perception Questionnaire (BIPQ) is a nine-item scale designed to assess the cognitive and emotional representations of illness. All of the items except the causal question (item 9) are rated using a 0 (most negative) to 10 (most positive) response scale from total score is calculated.
Absolute change in total IBS-SSS score and individual scores. | Baseline (Visit 2) to week 4 (call 1), to week 8 (call 2), and to week 12 (Visit 3)
  The IBS Symptom Severity Scale (IBS-SSS) contains 5 items. Each of the five questions generate a maximum score of 100 using prompted visual analogue scales. The maximum achievable score by an individual is 500.
Absolute change in the use of medications and treatments for bowel habits. | Baseline (2-week run-in period) to the last two weeks of intervention (week 11+12).
  Participants will report daily use of medications and treatments for bowel habits
Adverse Events by product causality | Baseline (Visit 2) to Week 12 (Visit 3)
  Proportion of AEs per group by product causality
Incidence of mild, moderate, and severe AEs | Baseline (Visit 2) to Week 12 (Visit 3)
  Incidence of mild, moderate, and severe AEs per group by product causality.
Severe Adverse Events (SAEs) by product causality | Baseline (Visit 2) to Week 12 (Visit 3)
  Incidence of SAEs per group by product causality
Vitals I | Baseline (Visit 2) to Week 12 (Visit 3)
  Change in systolic blood pressure (mmHg)
Vitals II | Baseline (Visit 2) to Week 12 (Visit 3)
  Change in diastolic blood pressure (mmHg)
Vitals III | Baseline (Visit 2) to Week 12 (Visit 3)
  Change heart rate (bpm)
Vitals IV | Baseline (Visit 2) to Week 12 (Visit 3)
  Change temperature (degrees ˚F)
Safety Labs | Baseline (Visit 2) to Week 12 (Visit 3)
  This outcome will report the incidence of 'out of range' blood safety parameters assessed from a standard safety chemistry panel and a standard safety hematology panel (Full Blood Count). 'Out of range' is determined based on clinically defined 'normal' ranges for each analyte. A higher incidence of 'out of range' blood safety parameters would be a worse safety outcome in this case.
Urinalysis (pH, protein, glucose, ketone, urobilinogen, bilirubin, blood, and nitrite). | Baseline (Visit 2) to Week 12 (Visit 3)
  This outcome will report the incidence of 'out of range' Urinalysis safety parameters (pH, protein, glucose, ketone, urobilinogen, bilirubin, blood, and nitrite). 'Out of range' is determined based on clinically defined 'normal' ranges for each analyte. A higher incidence of 'out of range' urinalysis safety parameters would be a worse safety outcome in this case.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Buckley, M.D., Principal Investigator — Atlantia Clinical Trials; Seema Mody, MSc, Study Director — DSM
Locations (1):
- Atlantia Clinical Trials Ltd, Cork, Cork/Munster, Ireland

IPD SHARING:
Plan to Share IPD: No